CLINICAL TRIAL: NCT06984731
Title: Clinical Trial Protocol for Safety and Efficacy of Transcatheter Ablation After Left Atrial Appendicular Occlusion With WATCHMAN FLX
Brief Title: The Safety and Efficacy of Radiofrequency Ablation After Left Atrial Appendage Occlusion.
Status: Recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-K080-01
Record Dates: First submitted 2025-04-22; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases; Arrhythmia
Keywords: Atrial Fibrillation (AF); Left Atrial Appendage closure with WATCHMAN device; Radiofrequency ablation
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Left Atrial Appendage Closure; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Patients who meet the diagnosis of non-valvular atrial fibrillation and plan to receive sequential treatment of WATCHMAN FLX left atrial appendage occlusion and transcatheter atrial fibrillation ablation.
  Interventions: Procedure: left atrial appendage closure; Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: left atrial appendage closure — Patients with atrial fibrillation underwent transcatheter radiofrequency cardiac ablation 1 month after left atrial appendage closure with WATCHMAN FLX
  Other Names: left atrial appendage closure with WATCHMAN FLX
Procedure: radiofrequency ablation — Patients with atrial fibrillation underwent transcatheter radiofrequency cardiac ablation 1 month after left atrial appendage closure with WATCHMAN FLX

SUMMARY:
Objective: To evaluate the safety and efficacy of transcatheter atrial fibrillation ablation 1 month after WATCHMAN FLX left atrial appendage closure in patients with nonvalvular atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common persistent arrhythmias in the clinic, and its incidence increases significantly with age, posing a serious threat to public health worldwide. One of the most serious complications in patients with atrial fibrillation is thromboembolic events, especially cardiogenic stroke. Cardiogenic stroke caused by atrial fibrillation accounts for 20%-30% of all stroke cases, and the mortality and disability rates of patients after stroke are significantly increased. Studies have shown that about 90% of the thrombus in patients with NVAF comes from the left atrial appendage (LAA). Therefore, isolating the left atrial appendage from the atrium to prevent stroke has become an important strategy in the management of patients with atrial fibrillation. This surgical method is called left atrial appendage occlusion (LAAO).

Moreover, both international and national guidelines for arrhythmia management indicate that rhythm control and stroke prevention are equally important for patients with atrial fibrillation. Although left atrial ear closure is effective in reducing the risk of stroke associated with atrial fibrillation, it does not address arrhythmia in patients. For heart rhythm control, catheter ablation is one of the most effective treatments available. It has been proven to significantly improve sinus rhythm maintenance and quality of life in patients with atrial fibrillation in several randomized controlled trials (RCTS). These studies suggest that catheter ablation is the preferred method for rhythm control in patients with paroxysmal AF, with better long-term results than medical treatment.

To comprehensively solve the problem of rhythm control and stroke prevention in patients with atrial fibrillation, the combination of catheter ablation and left atrial ear closure is a feasible and promising treatment strategy. Catheter ablation is designed to restore sinus rhythm by interfering with the triggering mechanism of atrial fibrillation, while left atrial appendage closure reduces stroke risk by isolating the main site of thrombosis. The combination of the two surgical methods not only improves the rate of sinus rhythm maintenance in patients but also significantly reduces the risk of stroke and all-cause death.

At present, the combined application of these two surgeries is gradually increasing in clinical practice. Some studies and expert consensus suggest that combined treatment goals can be achieved through "one-stop surgery" (performing both catheter ablation and left atrial appendage closure in one procedure) or phased surgery (performing one procedure before the other). However, there is no consensus on the optimal surgical sequence. Some studies have shown that "one-stop" surgery may shorten the length of hospital stay, and reduce surgical risks and patients' economic burden in the same period [13]. A phased procedure allows doctors to better evaluate the results after the initial surgery and reduce the overall surgical risk for the patient.

In the consensus of atrial fibrillation management experts in China in 2021, Category Ⅱb recommendation for "one-stop surgery" was proposed, suggesting that for some patients with nonvalvular atrial fibrillation who have indications of both catheter ablation and left atrial artery occlusion, it is reasonable to perform left atrial artery occlusion at the same time of catheter ablation. Despite this, there is currently a lack of trials to verify the safety and effectiveness of different surgical sequences.

Therefore, the purpose of this study was to evaluate the safety and effectiveness of transcranial atrial fibrillation ablation with WATCHMAN FLX 1 month after left atrial appendicular closure, to provide evidence-based medical evidence for optimizing the comprehensive management of patients with atrial fibrillation, and to further explore the optimal combined application strategy of the two surgical methods in patients with nonvalvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age, diagnosed with nonvalvular atrial fibrillation;
2. Meet the indications for receiving WATCHMAN FLX left atrial appendicular closure and transcatheter atrial fibrillation ablation;
3. Preoperative imaging evaluation showed that the anatomical structure of the left atrial appendage was suitable for implantation with the WATCHMAN FLX device;
4. The patient agrees to participate in the study and signs the informed consent.

Exclusion Criteria:

1. valvular heart disease or other structural heart disease that causes atrial fibrillation;
2. left auricular thrombus or acute thrombotic event was found before surgery;
3. Patients with severe bleeding tendency or recent major bleeding events (such as massive gastrointestinal bleeding, cerebral hemorrhage, etc.);
4. Patients who are unable to complete postoperative follow-up (such as life expectancy of less than 1 year or poor compliance);
5. Other serious diseases (such as liver and kidney failure, active infection, etc.) were found in preoperative examination;
6. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with symptomatic persistent atrial fibrillation, defined as: inability to spontaneously transition to sinus rhythm, lasting for more than 7 days, resistance or intolerance to at least Class I, II, or III antiarrhythmic drugs.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success at one year | one year
  The success rate of complete left atrial appendage closure within 12 months post-WATCHMAN FLX left atrial appendage occlusion surgery, as evaluated by contrast-enhanced computed tomography angiography (CTA) of the left atrial appendage.

SECONDARY OUTCOMES:
Rate of adverse events | one year
  The incidence of surgery-related complications and adverse events occurring within 30 days post-procedure following left atrial appendage occlusion and radiofrequency ablation was evaluated. This included the incidence of pericardial effusion, procedural access site complications, vascular complications, and infections.
  The incidence of surgery-related complications and adverse events within 12 months post-procedure was assessed. This encompassed severe bleeding (defined as bleeding requiring blood transfusion or surgical intervention), pericardial tamponade, systemic embolism (including ischemic stroke and other embolic events), occluder-associated thrombosis (DRT), new or enlarged residual shunt (PDL, defined as >5mm), postoperative acute left heart failure, and rehospitalization.
Arrhythmia recurrence during blanking period | one year
  The success rate of treatment within 3 months after radiofrequency ablation (early recurrence) : No recurrence of atrial arrhythmia ≥30 seconds;
Arrhythmia recurrence after blanking period | one year
  The success rate of treatment within 12 months after radiofrequency ablation (late recurrence) : There is no recurrence of atrial arrhythmia ≥30 seconds or more during the 4-12 months after the operation.
Incidence of stroke | one year
  Incidence of stroke within 12 months after left atrial appendage occlusion: No stroke occurred.
Quality of life changes at 12 months measured by AF Quality of Life Survey (AFEQT) | one year
  The improvement in quality of life between baseline and 12 months after the index ablation procedure or AAD measured by AF Quality of Life Survey (AFEQT) with the values ranging from 20 - 140 (higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT06984731/Prot_000.pdf